CLINICAL TRIAL: NCT03582163
Title: Longitudinal Outcomes of Deep Brain Stimulation in Parkinson's Disease
Brief Title: Longitudinal Outcomes of DBS in PD
Status: Terminated | Type: Observational
Why Stopped: Recruitment and enrollment were significantly slowed during the COVID-19 pandemic, and then research team effort shifted to another initiatives in interim.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Isaacs, Assistant Professor of Neurology, Vanderbilt University Medical Center
Other Study IDs: VUMCLODBSPD
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Longitudinal Outcomes; Subthalamic Nucleus; Globus Pallidus Interna
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- STN: Patients with Parkinson's disease who have undergone subthalamic nucleus (STN) DBS.
- GPi: Patients with Parkinson's disease who have undergone GPi (GPi) DBS.

SUMMARY:
Vanderbilt University Medical Center is one of the largest-volume DBS centers in the country. From 2007 through October 2017, 265 Parkinson's disease (PD) patients underwent deep brain stimulation (DBS), 168 of those implanted in subthalamic nucleus (STN) and 97 in globus pallidus interna (GPi). Pre-operatively, each patient is extensively evaluated with a battery of validated motor, cognitive, and mood instruments. This information is stored in RedCAP, a secure online database platform. In an attempt to capture longitudinal outcomes in this population of interest, we will recruit all PD patients two years or more status post DBS who are receiving regular care at Vanderbilt University Medical Center. Study participants will undergo a condensed evaluation of motor function (Unified Parkinson's Disease Rating Scale Part III), cognitive performance (Mini-Mental Status Examination), mood (Beck Depression Inventory), and quality of life (Parkinson's Disease Questionnaire-39). These results will be compared to baseline measures performed pre-operatively, allowing for assessment of interval change. STN and GPi DBS patients will be analyzed separately.

DETAILED DESCRIPTION:
Patients will be recruited from review of movement disorders neurologists' outpatient census. All patients with PD two or more years status post DBS will be contacted via phone and/or mailed letter. Any interested patient will be mailed or e-mailed (via RedCAP) a copy of the study informed consent form. Willing patients will present to the Vanderbilt Movement Disorders Clinic for an opportunity to inquire further about the study and sign the informed consent form in person.

Participants will have a single study visit, ideally coordinated with their regularly scheduled neurology follow-up. During the study visit, the following evaluations will be performed by a trained research assistant:

Video-recorded UPDRS III BDI MMSE PDQ-39 In addition, current PD medications and number of falls in the past 6 months will be recorded. Assessments will occur in the on-medication, on-DBS state.

The video-recorded UPDRS III will be reviewed and score at a subsequent date by a blinded rater (movement discord trained neurologist).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease
* status post deep brain stimulation (DBS) implantation in the subthalamic nucleus (STN) or globus pallidus interna (GPi) at Vanderbilt University Medical Center

Exclusion Criteria:

- unable to complete study assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The primary study base consists of all patients with Parkinson's disease 2 years or more status post DBS implantation at Vanderbilt University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale, Part III (UPDRS III) | at least 2 years
  Parkinson's disease motor assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No